CLINICAL TRIAL: NCT06739005
Title: artifiCiAl Intelligence Model for Evaluating the Surgical Techniques of caRdiAc Surgeons (CAMERA)
Brief Title: AI Model for Assessing Cardiac Surgeons' Techniques
Acronym: CAMERA
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Shengshou Hu, Academician of Chinese Academy of Engineering President, Fuwai Hospital Director, National Center for Cardiovascular Diseases Director, NCRC Director, State Key Laboratory of Cardiovascular Disease Chairman, China Heart Congress (CHC) Former President, China National Center for Cardiovascular Diseases
Other Study IDs: 2024-ZX070
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: CABG-patients; CABG; Cardiovascular Surgery; Surgeons; Artificial Intelligence (AI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study aims to investigate the use of artificial intelligence to analyze and evaluate the characteristics and proficiency of surgeons during vascular anastomosis in coronary artery bypass grafting (CABG) procedures. The main question it aims to answer is:

Consistency assessment between AI evaluation scores and human expert evaluation scores for surgeons during left anterior descending (LAD) artery anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing internal mammary artery-to-left anterior descending artery bypass grafting
* First-time recipient of isolated CABG surgery
* Signed written informed consent

Exclusion Criteria:

* Patients with acute coronary syndrome
* Patients with contraindications to coronary CT angiography or coronary angiography
* Patients with renal insufficiency or active liver disease, including those with persistently elevated serum transaminases of unknown cause or any serum transaminase levels exceeding three times the upper limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients who meet the inclusion criteria of being aged 18 years or older, undergoing their first isolated coronary artery bypass grafting (CABG) surgery using internal mammary artery-to-left anterior descending artery bypass grafting. All participants should signed written informed consent prior to inclusion in the study.
  Exclusion criteria include patients with acute coronary syndrome, contraindications to coronary CT angiography or coronary angiography, and those with renal insufficiency or active liver disease. Specifically, patients with persistently elevated serum transaminases of unknown cause or those with any serum transaminase levels exceeding three times the upper limit of normal will also be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 284 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Consistency assessment between AI surgical evaluation scores and human expert scores. | At the end of enrollment

SECONDARY OUTCOMES:
Intraoperative measurement of graft flow and flow resistance. | After enrollment
Characteristics of the surgeon's motion trajectory. | After enrollment
Consistency assessment between AI surgical evaluation scores levels and human expert scores levels. | After enrollment
  AI surgical evaluation scores levels were divided into the following 3 score levels: low, middle, high; human expert scores levels were divided into the following 3 score levels: low, middle, high.

OTHER OUTCOMES:
Graft patency at 1 year postoperatively. | At 1 year
Adverse cardiovascular events, such as myocardial infarction and stroke, within 6 months postoperatively. | At 6 months
Adverse cardiovascular events, such as myocardial infarction and stroke, within 12 months postoperatively. | At 12 months
Surgeon-level subgroup: age | Baseline
  Age subgroup is stratified into: <45, ≥45 years old
Surgeon-level subgroup: sex | Baseline
  Sex subgroup is stratified into: female, male
Surgeon-level subgroup: professional title | Baseline
  Professional title subgroup is stratified into: junior, associate, senior
Surgeon-level subgroup: annual surgery volume | Baseline
  Annual surgery volume subgroup is stratified by tertiles
Surgeon-level subgroup: total surgery volume | Baseline
  Total surgery volume subgroup is stratified by tertiles
Surgeon-level subgroup: annual CABG volume | Baseline
  Annual CABG volume subgroup is stratified by tertiles
Surgeon-level subgroup: total CABG volume | Baseline
  Total CABG volume subgroup is stratified by tertiles
Patient-level subgroup: age | Baseline
  Age subgroup is stratified into: <65, ≥65 years old
Patient-level subgroup: sex | Baseline
  Sex subgroup is stratified into: female, male
Patient-level subgroup: the severity of coronary artery disease | Baseline
  The severity of coronary artery disease is measured by SYNTAX score and is stratified into: <23, 23-32, >32

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, CAMS & PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yuan X, Liu F, Zhang L, Wang Y, Li J, Lei L, Gao S, Bao H, Yuan J, Zhang X, Feng W, Liu H, Zhao W, Hu S. Design and rationale of the artifiCiAl intelligence Model for Evaluating the surgical techniques of caRdiAc surgeons (CAMERA): a cohort study. BMJ Open. 2026 Feb 6;16(2):e106359. doi: 10.1136/bmjopen-2025-106359. PMID 41651534